CLINICAL TRIAL: NCT06963034
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Assess the Efficacy, Safety, and Tolerability of NBI-1117568 in Adults With Schizophrenia Who Warrant Inpatient Hospitalization
Brief Title: NBI-1117568-SCZ3029: Evaluation of NBI-1117568 in Inpatient Adults With Schizophrenia
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Neurocrine Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NBI-1117568-SCZ3029
Record Dates: First submitted 2025-04-30; First posted 2025-05-08 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NBI-1117568 (Experimental): Participants will receive NBI-1117568 once daily (QD) orally from Day 1 to Day 35 for a total of 5 weeks.
  Interventions: Drug: NBI-1117568
- Placebo (Placebo Comparator): Participants will receive matching placebo QD orally from Day 1 to Day 35 for a total of 5 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NBI-1117568 — NBI-1117568 will be administered per schedule specified in the arm description.
  Arms: NBI-1117568
Drug: Placebo — Placebo will be administered per schedule specified in the arm description.
  Arms: Placebo

SUMMARY:
The primary objective for this study is to evaluate the efficacy of NBI-1117568 compared with placebo on improving behavioral and psychological symptoms of schizophrenia in adults.

ELIGIBILITY:
Key Inclusion Criteria:

* Participant has a primary diagnosis of schizophrenia
* Participant is experiencing an acute exacerbation or relapse of symptoms and currently warrants hospitalization.
* Participants taking prohibited medications, including antipsychotics, must discontinue before study participation
* Participant is willing and able to remain in an inpatient setting for the study duration, follow instructions, and comply with the protocol requirements

Key Exclusion Criteria:

* Participant has known hypersensitivity to any component of the formulation of NBI-1117568.
* Participant has an unstable or poorly controlled medical condition or chronic disease
* Participant is considered by the investigator to be at imminent risk of suicide or injury to self or others
* Participant has a diagnosis of moderate or severe substance use disorder (with the exception of nicotine or caffeine dependence) within 6 months prior to screening
* Participant has a positive alcohol test or drug screen for disallowed substances
* Participants have a history of poor or suspected poor compliance in clinical research studies and/or in the investigator's opinion, the participant is not capable of adhering to the protocol requirements.

Note: Other protocol-specified inclusion/exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 284 (Estimated)
Dates: Start 2025-05-08 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Total Score at Week 5 | Baseline, Week 5

SECONDARY OUTCOMES:
Change From Baseline in Clinical Global Impression - Severity (CGI-S) Score at Week 5 | Baseline, Week 5

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Lead, Study Director — Neurocrine Biosciences
Locations (20):
- United States (20):
  - Neurocrine Clinical Site, Little Rock, Arkansas
  - Neurocrine Clinical Site, Anaheim, California
  - Neurocrine Clinical Site, Pico Rivera, California
  - Neurocrine Clinical Site, San Diego, California
  - Neurocrine Clinical Site, Sherman Oaks, California
  - Neurocrine Clinical Site, Torrance, California
  - Neurocrine Clinical Site, Hollywood, Florida
  - Neurocrine Clinical Site, Miami Lakes, Florida
  - Neurocrine Clinical Site, Atlanta, Georgia
  - Neurocrine Clinical Site, Decatur, Georgia
  - Neurocrine Clinical Site, Peachtree Corners, Georgia
  - Neurocrine Clinical Site, Chicago, Illinois
  - Neurocrine Clinical Site, Gaithersburg, Maryland
  - Neurocrine Clinical Site, Watertown, Massachusetts
  - Neurocrine Clinical Site, Marlton, New Jersey
  - Neurocrine Clinical Site, Staten Island, New York
  - Neurocrine Clinical Site, The Bronx, New York
  - Neurocrine Clinical Site, Austin, Texas
  - Neurocrine Clinical Site, DeSoto, Texas
  - Neurocrine Clinical Site, Houston, Texas